CLINICAL TRIAL: NCT04207385
Title: Accurate Clinical Study of Medication in Patients With Depression Via Pharmacogenomics (PGx) and Therapeutic Drug Monitoring (TDM) of Venlafaxine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20192104-X-1
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-11

CONDITIONS: Depression
Keywords: pharmacogenomics; PGx; therapeutic drug monitoring; TDM; Venlafaxine; depression
MeSH Terms: conditions — Depression | interventions — Pharmacogenomic Testing; Drug Monitoring; Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- A group: Routine treatment group (Active Comparator): Routine dosage of venlafaxine during the first 4 weeks.
  Interventions: Drug: Venlafaxine
- B group: PGx-guided group (Experimental): The PGx test results guide the dosage of venlafaxine during the first 4 weeks.
  Interventions: Diagnostic Test: pharmacogenomics; Drug: Venlafaxine
- C group: Routine PGx-guided group (Active Comparator): The PGx test results guide the dosage of venlafaxine between 4th and 8th weeks.
  Interventions: Diagnostic Test: pharmacogenomics; Drug: Venlafaxine
- D group: The combination of PGx and TDM group (Active Comparator): The PGx and TDM test results guide the dosage of venlafaxine between 4th and 8th weeks.
  Interventions: Diagnostic Test: pharmacogenomics; Diagnostic Test: pharmacogenomics & therapeutic drug monitoring; Drug: Venlafaxine

INTERVENTIONS:
Diagnostic Test: pharmacogenomics — pharmacogenomics
  Arms: B group: PGx-guided group; C group: Routine PGx-guided group; D group: The combination of PGx and TDM group
Diagnostic Test: pharmacogenomics & therapeutic drug monitoring — pharmacogenomics & therapeutic drug monitoring
  Arms: D group: The combination of PGx and TDM group
Drug: Venlafaxine — Venlafaxine hydrochloride sustained-release capsules 75mg x 14 tablets x 1 case 75-225mg/morning

SUMMARY:
This study evaluates the efficacy of PGx-guided medication in patients with depression treated with Venlafaxine and the efficacy of the combination of PGx and TDM in patients with depression treated with Venlafaxine. Half of participants will receive PGx-guided treatment, while the other half will receive routine treatment. After the 8th week, the PGx-guided treatment group would be randomly divided into two groups. Of which, half of participants will receive the combination of PGx and TDM, and the other half will receive PGx -guided medication only.

DETAILED DESCRIPTION:
The current clinical medication is based on "Trial and Error", while the traditional medication is mainly based on experience. The study mainly optimizes the treatment path from two perspectives: to help clinicians select drugs accurately through the detection of PGx; to help clinicians monitor the whole process of drug use through TDM and adjust the dosage in time to achieve better treatment.

PGx tests take the information of metabolic, transporting and target genetic factors into account comprehensively. Furthermore, clinical effects depend on blood concentration rather than dose concentration. TDM aims to monitor blood concentration, which is related to drug efficacy and toxicity.

Venlafaxine is an antidepressant drugs of the 5-hydroxytryptamine selective seratonin re-uptake inhibitors (SSRIs), which has been approved by FDA for the treatment of depressive disorders, depressive disorders with anxiety symptoms, generalized anxiety disorders and social anxiety disorders since 1994.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endogenous depression, with any of the following 4 symptoms: ① Interest Loss; ② Hypothymia; ③ Early awakening; ④ Serious in the morning and relieved at night; ⑤ Hysteresis or agitation of movement of Spirit; ⑥ Appetite loss; ⑦ Weight loss; ⑧ Loss of libido;
* Scores of 17 items in Hamilton Depression Scale (HAM-D17): over 17 points;
* First-episode patients or relapsed patients without taking any antidepressant drugs in the recent 3 months;
* No significant abnormalities are shown in physical examination (temperature, pulse, blood pressure, head and neck, chest and abdomen).
* No obvious abnormalities in laboratory examination (Thyroid Function).
* Informed patient consent.

Exclusion Criteria:

* Those diagnosed with mental disorders other than major depressive disorders (with the exception of combination of anxiety disorders); non-endogenous depressive disorders;
* Patients with stroke, brain tumor and other brain organic diseases;
* Patients receiving combined drugs (but there is no need to exclude patients receving drugs against sleep disorders, such as Eszopiclone, alprazolam or estazolam);
* History of drug allergy;
* Pregnant and lying-in women;
* Patients with serious suicidal tendencies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
Score reduction rate of Hamilton Depression Rating Scale | 3 days
  Reduction Rate=[(total score before treatment-total score after treatment)/total score before treatment] *100%
  * Healed: reduction rate ≥ 75%;
    * Significant Effective: reduction rate≥50％and <75％; ③Effective: reduction rate≥25％ and <50％; ④Invalid: Reduction rate < 25%

CONTACTS AND LOCATIONS:
Overall Officials: Huaning Wang, Study Chair — Deputy Chief Physician; Ping Zhou, Principal Investigator — Attending Physician; Yihuan Chen, Principal Investigator — Attending Physician; Huizhen Lu, Principal Investigator — Resident Physician; Qinghong Yan, Principal Investigator — Nurse
Locations (1):
- Xijing Hospital, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No